CLINICAL TRIAL: NCT00712985
Title: Single Dosing of Zoledronic Acid in Cancer Therapy Induced Bone Loss (CTIBL)
Acronym: CTIBL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Allan Lipton, MD, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CZOL446H US113
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Results first posted 2014-04-24 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-03

CONDITIONS: Breast Cancer
Keywords: Breast cancer; aromatase inhibitors
MeSH Terms: conditions — Breast Neoplasms | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Zometa (Zoledronic Acid) X 1 dose (Experimental): Zometa (Zoledronic Acid) 5 mg IV X 1 dose
  Interventions: Drug: Zometa

INTERVENTIONS:
Drug: Zometa — Zometa (Zoledronic Acid) 5 mg IV over 15 minutes in a one time dose
  Other Names: Zoledronic Acid

SUMMARY:
The purpose of this research is to establish if a once a year dose of Zoledronic Acid is sufficient to suppress and maintain urine and serum bone density markers (NTx) and serum CTx within normal range at 12 months post-dosing in postmenopausal early breast cancer patients receiving additional treatment with non-steroidal aromatase inhibitors.

DETAILED DESCRIPTION:
Bone metastases are frequently one of the first signs of disseminated disease in cancer patients. Skeletal complications due to metastatic disease include (severe) bone pain, spinal cord compromise, pathological fractures, and hypercalcemia.

Zoledronic acid is a member of a class of compounds known as bisphosphonates. Bisphosphonates are effective inhibitors of osteoclastic bone resorption and have demonstrated therapeutic efficacy in the treatments of hypercalcemia of malignancy, lytic bone disease associated with multiple myeloma, and mixed lytic and blastic bone metastases associated with breast cancer. The precise mechanism by which bisphosphonates inhibit osteoclast function is not fully understood, but may include a direct toxic effect on mature osteoclasts, an inhibition of osteoclast production from precursor cells, and an impairment of osteoclast chemotaxis to sites of active bone resorption. Osteoclasts are specialized bone cells which erode mineralized bone by secreting acids and lysosomal enzymes. In normal bone remodeling, osteoclastic bone resorption is coupled to and is in equilibrium with osteoblastic bone formation. The lytic bone destruction associated with malignant bone metastases develops because tumor cells synthesize and release soluble factors that stimulate osteoclasts to resorb bone. The osteoclastic activating factors released by tumor cells include parathyroid hormone-related peptide (PTHrP), growth factors, and cytokines. The malignant activation of osteoclasts results in a disruption of normal bone remodeling wherein the equilibrium between bone resorption and bone formation is shifted toward increased bone resorption. This relative increase in osteoclastic bone resorption results in a net loss of bone. Thus, the predominant role of the osteoclast in the pathogenesis of bone destruction and the inhibitory effects of bisphosphonates on osteoclast function have formed the rationale for the use of bisphosphonates in the treatment of osteolytic bone metastases. The common role, regardless of tumor type, of the osteoclast as the mediator of bone destruction in metastatic skeletal disease is indicated by the inhibitory effects of bisphosphonates on tumor-induced osteolysis in animal models utilizing various malignant cell lines and the effectiveness of bisphosphonates in the therapy of tumor-induced hypercalcemia arising from any type of cancer. Moreover, recent studies have specifically shown that therapy with the bisphosphonate pamidronate (Aredia) combined with antineoplastic therapy significantly reduces the proportion of patients having skeletal complications due to the lytic bone disease associated with multiple myeloma and breast cancer compared to antineoplastic therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with Stage I, II or IIIa breast cancer being treated with a non-steroidal Aromatase Inhibitor (AI) .Negative bone scan (no bone metastases).
* Calculated creatinine clearance > 40 ml/min
* Documented T score of less than or equal to -1.5 on Dual Energy X-ray Absorptiionmetry (DXA) scan at the lumbar spine or femoral neck within 3 months prior to screening.
* Urine NTx > 50 nano moles(nM)based on second morning void.
* Signed informed consent.
* Ambulatory patients at least 18 years of age.
* Eastern Cooperative Oncology Group (ECOG)0-2.
* Ability to comply with trial requirements.

Exclusion Criteria:

* Bone Metastases.
* Any woman of child bearing potential.
* Patients with fractures occurring within three months prior to randomization. - Greater than a 2+ protein on urine dipstick without evidence of contamination or bacteriuria (may be repeated one time, at least a day apart).
* Calculated creatinine clearance less than 30 mL/min at screening.
* Serum calcium > 2.75 mmol/L (11.0 mg/dL) or < 2.00 mmol/L (8.0 mg/dL).
* Liver Function tests (LFT)> 2.0 x upper limit of normal (ULN).
* Serum alkaline phosphatase > 1.5 x ULN. History of hypersensitivity to bisphosphonates.
* Evidence of vitamin D deficiency (serum 25-(OH) D of less than 15 ng/ml).
* History of uveitis or iritis, except when secondary to trauma, and must have resolved > 2 years prior to entry.
* A history of invasive malignancy of any organ system, treated or untreated, within the past 12 months prior to screening; excluding, basal cell or squamous cell carcinoma of the skin, colonic polyps with non-invasive malignancy which have been removed, Ductal Carcinoma in-situ (DCIS) that has been surgically removed, and Carcinoma in-situ (CIS) of the uterine cervix that has been surgically removed.
* Previous major solid organ transplant recipient or on a transplant waiting list.
* Treatment with any investigational drug within 30 days prior to randomization.
* History of hyperparathyroidism, hypoparathyroidism, Osteogenesis imperfecta, Paget's disease or any metabolic bone disease other than osteoporosis.
* Any medical condition which would interfere with the action of the study drug or limit life expectancy to less than 6 months.
* Any medical or psychiatric condition which, in the opinion of the investigator, would preclude the participant from adhering to the protocol or completing the trial.
* Prior treatment with IV bisphosphonates within the last 2 years.
* Previous use of oral bisphosphonates within the past 2 years (unless used for less than 8 weeks*). *NOTE: If used less than 8 weeks, the washout period is 6 months.
* Treatment with raloxifene, calcitonin, tibolone or hormone replacement therapy. The washout period for these medications is 6 months prior to randomization.
* Any treatment with strontium ranelate, samarium, sodium fluoride or parathyroid hormone.
* Use of systemic high dose corticosteroids at an average dose of > 7.5 mg per day of oral prednisone or equivalent for a period of three months or more prior to screening.
* Known hypersensitivity to zoledronic acid or other bisphosphonates.
* Current active dental problems including infection of the teeth or jawbone (maxilla or mandibular); dental or fixture trauma, or a current or prior diagnosis of osteonecrosis of the jaw (ONJ), of exposed bone in the mouth, or of slow healing after dental procedures.
* Recent (within 6 weeks) or planned dental or jaw surgery (e.g.. extraction, implants).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2005-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allan Lipton, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Baum M, Budzar AU, Cuzick J, Forbes J, Houghton JH, Klijn JG, Sahmoud T; ATAC Trialists' Group. Anastrozole alone or in combination with tamoxifen versus tamoxifen alone for adjuvant treatment of postmenopausal women with early breast cancer: first results of the ATAC randomised trial. Lancet. 2002 Jun 22;359(9324):2131-9. doi: 10.1016/s0140-6736(02)09088-8. PMID 12090977
- [Background] Goss PE, Ingle JN, Martino S, Robert NJ, Muss HB, Piccart MJ, Castiglione M, Tu D, Shepherd LE, Pritchard KI, Livingston RB, Davidson NE, Norton L, Perez EA, Abrams JS, Therasse P, Palmer MJ, Pater JL. A randomized trial of letrozole in postmenopausal women after five years of tamoxifen therapy for early-stage breast cancer. N Engl J Med. 2003 Nov 6;349(19):1793-802. doi: 10.1056/NEJMoa032312. Epub 2003 Oct 9. PMID 14551341
- [Background] Coombes RC, Hall E, Gibson LJ, Paridaens R, Jassem J, Delozier T, Jones SE, Alvarez I, Bertelli G, Ortmann O, Coates AS, Bajetta E, Dodwell D, Coleman RE, Fallowfield LJ, Mickiewicz E, Andersen J, Lonning PE, Cocconi G, Stewart A, Stuart N, Snowdon CF, Carpentieri M, Massimini G, Bliss JM, van de Velde C; Intergroup Exemestane Study. A randomized trial of exemestane after two to three years of tamoxifen therapy in postmenopausal women with primary breast cancer. N Engl J Med. 2004 Mar 11;350(11):1081-92. doi: 10.1056/NEJMoa040331. PMID 15014181
- [Background] BIG 1-98 Collaborative Group. Letrozole versus tamoxifen as adjuvant endocrine therapy for postmenopausal women with receptor-positive breast cancer. BIG 1-98: a prospective randomized double-blind phase III study. Breast. 2005;14:Suppl 1:S3. Abstract.
- [Background] Walsh PC. Intravenous zoledronic acid in postmenopausal women with low bone mineral density. J Urol. 2002 Oct;168(4 Pt 1):1643. No abstract available. PMID 12356057
- [Background] Smith MR, Eastham J, Gleason DM, Shasha D, Tchekmedyian S, Zinner N. Randomized controlled trial of zoledronic acid to prevent bone loss in men receiving androgen deprivation therapy for nonmetastatic prostate cancer. J Urol. 2003 Jun;169(6):2008-12. doi: 10.1097/01.ju.0000063820.94994.95. PMID 12771706

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was from 1/10/2007 for first patient consented to 12/29/2009 last patient consented. The patients were all seen in the Milton S. Hershey Medical Center Oncology clinic & were treated from first patient Day 1 of 1/16/2007 to last patient month 12 of 2/01/2011.
Pre-assignment Details: Following consent, this trial only had 1 arm & all patients were given a one time dose of Zoledronic Acid 5 mg IV. All 17 patients were then followed for 12 months from day 1 & their urine & serum were collected in order to evaluate the urine N-telopeptide (NTx) & serum NTx & C-telopeptide (CTx) levels.
Groups:
- Zoledronic Acid 5 mg IV: Zometa (Zoledronic Acid) 5 mg IV given over 15 minutes as a one time dose. Follow-up at month 1 & every 2 months to month 12 for serum & urine markers of bone destruction (NTx & CTx).
Period: Overall Study
Arm/Group | Zoledronic Acid 5 mg IV
Started | 18
Completed | 13
Not Completed | 5
Not completed — 1 withdrew prior to start of drug | 1
Not completed — 1 patient moved out of state | 1
Not completed — Lack of Efficacy | 3

BASELINE CHARACTERISTICS:
Population: 18 patients signed consent & 1 withdrew due to family not wishing her to continue with trial.
Arm/Group | Zoledronic Acid 5 mg IV
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (9.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Urine and Serum NTx and Serum CTx Within Normal Range at 12 Months
Description: 17 women with early breast cancer receiving adjuvant Aromatase Inhibitor (AI) therapy were treated with a single 5 mg IV dose of zoledronic acid. Urine and serum NTx and serum CTx were measured at baseline and month 12.
Time Frame: One year
Measure: Number; unit: participants
Arm/Group | Zoledronic Acid 5 mg IV
Number analyzed (Participants) | 13
participants | 13

ADVERSE EVENTS:
Time Frame: Monthly for 1 year
Arm/Group | Zoledronic Acid 5 mg IV
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

LIMITATIONS AND CAVEATS:
18 patients were able to be enrolled in this trial & only 13 were able to be analyzed. This was an insufficient number to analyze/interpret data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No